CLINICAL TRIAL: NCT03710304
Title: The Effect of IV Tranexamic Acid Plus Buccal Misoprostol on Blood Loss During and After Cesarean Delivery: a Randomized Controlled Trial
Brief Title: Tranexamic Acid Plus Buccal Misoprostol on Blood Loss During and After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/173/7/18
Record Dates: First submitted 2018-10-13; First posted 2018-10-18 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; tranexamic acid; postpartum hemorrhage; buccal misoprostol
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Tranexamic Acid; Misoprostol

STUDY DESIGN:
Intervention Model Description: participants will be randomized via a computer-generated random number sequence into one of two groups: one group received a pre-prepared sealed and opaque packet containing 400 μg of misoprostol (2 tablets of 200 μg), 2 ampoules of TA (1 gm for infusion) and separate placebo ampoule (distilled water). The other group received similar packets containing two placebo tablets, two placebo ampoules (distilled water) and separate 2 ampoules of oxytocin (syntocinon; 10 IU in each ampoule for infusion) for slow intravenous injection. The misoprostol and placebo tablets were similar in size, shape, and color, and ampoules of oxytocin was also similar to placebo. Randomization was done by the resident doctors immediately before transfer to theater, whereas preparation of packets and confidential record maintenance was done by the labor room nursing staff.
  Study drug administration
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin (Active Comparator): 20 IU oxytocin ampoules in 500 mL of intravenous solution infusion over 15 min after delivery of the baby.plus 2tab placebo buccal(ranitidine) plus 110 ml saline iv
  Interventions: Drug: Oxytocin
- Tranexamic acid plus misoprostol (Active Comparator): 400 μg misoprostol (2 tablets of 200 μg) or two placebo tablets were given buccally after spinal anesthesia and few minutes before skin incision; then 1 gm TA will be diluted in 100 mL normal saline and administered slowly (over 30-60 s) intravenously by the anesthetist before skin incision, plus 500 ml normal saline intravenous solution infusion over 15 min after delivery of the baby
  Interventions: Drug: Tranexamic acid plus misoprostol; Drug: misoprostol

INTERVENTIONS:
Drug: Oxytocin — 20 IU oxytocin or placebo ampoules in 500 mL of intravenous solution infusion over 15 min after delivery of the baby.plus 2tab placebo buccal plus 110 ml saline by slow infusion
  Other Names: Active Comparator
  Arms: oxytocin
Drug: Tranexamic acid plus misoprostol — 1 gm TA or separate placebo will be diluted in 100 mL normal saline and administered slowly (over 30-60 s) intravenously by the anesthetist before skin incision,
  Other Names: Active Comparator
  Arms: Tranexamic acid plus misoprostol
Drug: misoprostol — 400 μg misoprostol (2 tablets of 200 μg) will be give buccally after spinal anesthesia and few minutes before skin incision;
  Other Names: Active Comparator
  Arms: Tranexamic acid plus misoprostol

SUMMARY:
Postpartum hemorrhage (PPH) is potentially life-threatening and is a significant contributor to maternal mortality and morbidity especially in developing countries.

The risk of PPH is much higher for women undergoing cesarean delivery (CD). In the majority of cases, uterine atony is responsible for the occurrence of excessive bleeding during or following childbirth.

The Millennium Development Goal of reducing the maternal mortality ratio by 75 % by 2015 will remain beyond our reach unless we prioritize the prevention and treatment of PPH in low-resource countries.

Consequently, the administration of uterotonic drugs during cesarean section (CS) and in the third stage of labor for vaginal delivery has become essential to diminish the risk of PPH and improve maternal safety.

Oxytocin is regarded as the gold standard uterotonic agent but only has a half-life of 4-10 min; therefore, at cesarean section oxytocin must be administered as a continuous intravenous infusion to attain sustained uterotonic activity throughout the surgical procedure and immediate postpartum period.

Misoprostol is a prostaglandin E1 analog proven in several randomized controlled trials to be effective in preventing PPH because of its strong uterotonic effects. In addition, misoprostol is inexpensive, stable at room temperature, and easy to administer.

Misoprostol has been broadly studied in the prevention and treatment of PPH after vaginal delivery; however, its use in conjunction with CD has not been investigated as much.

The buccal route is recognized as having the greatest benefit due to its rapid uptake, long-acting effect, and greatest bioavailability compared with other routes of misoprostol administration.

Tranexamic acid(TA) is a synthetic analog of the amino acid lysine,10 as an antifibrinolytic agent it has roughly eight times the antifibrinolytic activity of an older analog; ε-aminocaproic acid.

The aim of this study was to compare the effectiveness of combined buccal misoprostol and intravenous TA with intravenous oxytocin for the prevention of PPH in patients with risk factors during cesarean section.

DETAILED DESCRIPTION:
Eligible and consenting participants were randomized via a computer-generated random number sequence into one of two groups: one group received a pre-prepared sealed and opaque packet containing 400 μg of misoprostol (2 tablets of 200 μg), 2 ampoules of TA (1 gm for infusion) and separate placebo ampoule (distilled water). The other group received similar packets containing two placebo tablets, two placebo ampoules (distilled water) and separate 2 ampoules of oxytocin (10 IU in each ampoule for infusion) for slow intravenous injection. The misoprostol and placebo tablets were similar in size, shape, and color, and ampoules of oxytocin will be also similar to placebo. Randomization was done by the investigator immediately before transfer to the theater, whereas the preparation of packets and confidential record maintenance was done by the labor room nursing staff.

Study drug administration 400 μg misoprostol (2 tablets of 200 μg) or two placebo tablets were given buccally after spinal anesthesia and few minutes before skin incision; then 1 gm TA or separate placebo will be diluted in 100 mL normal saline and administered slowly (over 30-60 s) intravenously before skin incision, in group 2 20 IU oxytocin or placebo ampoules in 500 mL of intravenous solution infusion over 15 min after delivery of baby.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for an elective cesarean section with risk factors for atonic PPH

Exclusion Criteria:

* Patients with a cardiac, hepatic, renal or thromboembolic disease
* patients had an allergy to tranexamic acid
* suspected coagulopathy
* history of coronary artery disease or hypertension
* patient refuses to participate

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — patients scheduled for an elective cd with risk factors for atonic PPH during cesarean section
Enrollment: 400 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
number of participant required of additional pharmacological uterotonic. | 24 hours post operative
  the number of participant need for extra uterotonic drug

SECONDARY OUTCOMES:
difference between preoperative and postoperative hemoglobin | 24 hours post operative
  compare of hemoglobin in gm/dl preoperative and 24 hours post operative
intraoperative blood loss | during the operation
  amount of blood loss during the operation
post operative blood loss | 24 hours post operative
  amount of blood loss from the end of operation till 24 hours post operative

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No